CLINICAL TRIAL: NCT03126006
Title: The Effect of Non-surgical Periodontal Therapy on Adverse Birth Outcomes: A Randomized Controlled Trial
Brief Title: The Effect of Non-surgical Periodontal Therapy on Adverse Birth Outcomes Randomized Controlled Trial
Acronym: NSPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Farhan Raza Khan, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3232-CHS-ERC-14
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Birth Weight; Birth, Preterm
MeSH Terms: conditions — Birth Weight; Premature Birth | interventions — Oral Hygiene; Tooth Exfoliation; Dental Scaling; Periodontal Debridement; Hygiene

STUDY DESIGN:
Intervention Model Description: It's an assessor blinded, parallel group, randomized controlled trial aimed at determining the superiority of non-surgical periodontal therapy over no dental treatment among pregnant women.
  The main objective of this trial is to determine whether the provision of NSPT to pregnant women with periodontitis is effective in reducing the incidence of low birth weight, preterm birth and still birth when compared to the pregnant women who were subjected to no NSPT. Outcomes of interest are pre-term birth (<37 weeks) gestation, low birth weight (<2500g) or still birth with either one occurring being considered as a positive outcome.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSPT plus oral hygiene (Experimental): It includes pregnant women (with periodontal disease) who will be subjected to one episode of non-surgical periodontal therapy under local anesthesia during pregnancy. they will receive oral hygiene instruction also.
  Interventions: Procedure: NSPT plus oral hygiene
- Oral hygiene alone (Other): It includes pregnant women (with periodontal disease) who will not be given any mechanical treatment such as non-surgical periodontal therapy during pregnancy. However, oral hygiene instructions will be given.
  Interventions: Other: Oral hygiene alone

INTERVENTIONS:
Procedure: NSPT plus oral hygiene — Non-surgical periodontal therapy under local anesthesia to remove plaque and calculus
  Other Names: scaling, dental scaling, de-scaling; periodontal prophylaxis, periodontal debridement
  Arms: NSPT plus oral hygiene
Other: Oral hygiene alone — It includes pregnant women (with periodontal disease) who will not be given any mechanical treatment such as non-surgical periodontal therapy during pregnancy. However, oral hygiene instructions will be given.
  Arms: Oral hygiene alone

SUMMARY:
The main objective of this study is to determine whether the provision of non-surgical periodontal therapy to pregnant women with periodontitis is effective in reducing the incidence of low birth weight, preterm birth and still birth when compared to pregnant women with periodontitis but who will be provided with oral hygiene instructions alone.

DETAILED DESCRIPTION:
Approximately two-thirds of pregnant Pakistani women suffer from periodontal disease a common inflammatory disease of the soft tissues surrounding the tooth. It was demonstrated that periodontitis among pregnant women is significantly associated with preterm birth and low birth weight. Pakistan has a high prevalence of these adverse birth outcomes therefore; identifying an intervention is of prime importance and may have social and economic benefits.

Non-surgical periodontal therapy is affordable and amenable to people and thus seems to be an intervention which may prove to be of benefit in a population where the dental services are available. It has been recommended in systematic reviews and Meta analysis that Randomized Controlled Trials are now required to establish whether the removal of inflammatory factors by scaling and root planning are effective in reducing adverse pregnancy outcomes such as preterm birth and low birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman presenting to the Obstetric clinic at the Aga Khan Hospital for Women, Karimabad or the Aga Khan Hospital for Women and Children, Kharadar.
* Participant should be between the ages of 18 and 35 years
* Exhibiting at least 2 sites with 2mm or more periodontal probing depth.
* Planning to deliver the baby at the above mentioned facilities so that the outcome can be observed and measured.
* Singleton pregnancy.
* Willing to get NSPT done between 20 to 28 weeks of gestation.
* At least 20 teeth present in the mouth so that periodontal scoring could be done.

Exclusion Criteria:

* Tobacco or alcohol use.
* Genitourinary tract infection or any systemic infection.
* Obstetric disorders such as gestational diabetes or placenta previa or pre-eclampsia or eclampsia etc.
* Chronic disease such as diabetes or blood pressure.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women only
Enrollment: 115 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Premature birth | To be assessed at birth
  less than 37 weeks

SECONDARY OUTCOMES:
Birth weight | To be assessed at birth
  less than 2500grams
Still birth | To be assessed at birth
  To be assessed by the birth attendant/ Obgyne

CONTACTS AND LOCATIONS:
Overall Officials: Zaubina U Kazi, BDS, MSc, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No